CLINICAL TRIAL: NCT02069366
Title: Cannabinoid Control of Fear Extinction Neural Circuits in Post-traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Christine Rabinak, PhD, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1K01MH101123-01A1 (NIH)
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Results first posted 2022-09-09 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Post-Traumatic Stress Disorders; Dronabinol; Extinction; fMRI
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Dronabinol; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): In a randomized, double-blind, placebo-controlled, between-subjects design, we will administer a one-time oral dose of dronabinol (7.5mg) or placebo (PBO) approximately two hours prior to fMRI scanning and task performance in 40 patients with PTSD, 40 trauma-exposed controls without PTSD (TEC), and 40 non-exposed healthy controls (HC).
  Within each of the three groups half of the participants will receive dronabinol and the other half will received placebo to create the following 6 groups:
  1. PTSD-dronabinol (20)
  2. PTSD-placebo (20)
  3. TEC-dronabinol (20)
  4. TEC-placebo (20)
  5. HC-dronabinol (20)
  6. HC-placebo (20)
  Interventions: Drug: Placebo
- Dronabinol (Active Comparator): In a randomized, double-blind, placebo-controlled, between-subjects design, we will administer a one-time oral dose of dronabinol (7.5mg) or placebo (PBO) approximately two hours prior to fMRI scanning and task performance in 40 patients with PTSD, 40 trauma-exposed controls without PTSD (TEC), and 40 non-exposed healthy controls (HC).
  Within each of the three groups half of the participants will receive dronabinol and the other half will received placebo to create the following 6 groups:
  1. PTSD-dronabinol (20)
  2. PTSD-placebo (20)
  3. TEC-dronabinol (20)
  4. TEC-placebo (20)
  5. HC-dronabinol (20)
  6. HC-placebo (20)
  Interventions: Drug: Dronabinol

INTERVENTIONS:
Drug: Dronabinol — Dronabinol (7.5mg) is administered only once (approximately 120 min prior to fMRI scanning in Visit 3) by the oral route and is placed in opaque capsules with dextrose filler. Half of the participants in each diagnostic group [HC = 20; PTSD = 20; TEC = 20] will receive dronabinol.
  Other Names: Marinol
  Arms: Dronabinol
Drug: Placebo — Placebo is administered only once (approximately 120 min prior to fMRI scanning in Visit 3) by the oral route and contains only dextrose in opaque capsules. Half of the participants in each diagnostic group [HC = 20; PTSD = 20; TEC = 20] will receive placebo.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The goal of this study is to look at how a type of drug called cannabinoids are related to the processing of fear signals, the experience of emotions and fear, and the pattern of activity in the brain that is involved in these processes and how this relates to the development of post-traumatic stress disorder (PTSD). PTSD is an anxiety disorder that occurs after experiencing a traumatic event(s) and is characterized by unwanted memories of the trauma(s) through flashbacks or nightmares, avoidance of situations that remind the person of the event, difficulty experiencing emotions, loss of interest in activities the person used to enjoy, and increased arousal, such as difficulty falling asleep or staying asleep, anger and hypervigilance. The information gained from this study could lead to the development of new treatments for persons who suffer from anxiety or fear-based disorders.

DETAILED DESCRIPTION:
The total time that for each participant involved in this study is 4 visits, as outlined below:

Visit 1: Questionnaires, Screening, and Orientation: During this visit the potential participant will learn about the study procedures, sign the informed consent documents, and fill out a packet of forms that ask about his or her race and ethnic background, use of drugs and alcohol and physical and mental health.

Visit 2: Behavioral Tests: During this visit the participant will complete several computer tasks, and the study staff will be measuring reaction time and psychophysiological measures.The tasks that the participant will perform will show three different images and an aversive stimulus (e.g. loud burst of noise or mild wrist shock) may follow one image most of the time, while the other images may never be followed by a noise or mild wrist shock. The participant will need to try to predict whether the aversive cue will occur or not based on which image is shown and will be asked to repeatedly rate on a scale how likely it is that he or she thinks a noise/shock will occur after each image. Lastly, during the session the participant will also be asked to report his or her level of anxiety on a scale from 0 to 100.

Visit 3: Behavioral Tests with Drug or Placebo and MRI scan: For safety reasons participant will not be allowed to take any drugs for at least 24 hours before this visit, and should not use marijuana for at least 2 weeks before. Participants will be required to pass a urine drug test (and pregnancy test for women) and breathalyzer test before being allowed to continue with this visit. The participant will also not be allowed to drive himself or herself home from this visit, so he or she should arrange a friend or family member to pick him or her up or a taxi can be called by our research staff.

The participant will view the same images he or she did on the previous day (Visit 2), and may experience the same aversive stimulus as during Visit 2. The participant will again be asked to rate how much he or she expects to experience the aversive stimulus after each image and he or she will also be asked to report his or her level of anxiety on a scale from 0 to 100. However, about 2 hours before the task begins, the participant will be asked to swallow a capsule containing either a marijuana-like drug (Dronabinol) or a placebo (sugar pill). Dronabinol is a Food & Drug Administration (FDA) approved drug and the dose (7.5mg; one time) is unlikely to have any effects that last beyond the duration of the study visit. About every 30 minutes after taking the pill, the participant will fill out some questionnaires about mood and how he or she is feeling at the moment.

Visit 4: Behavioral Tests and MRI scan: This visit will be very similar to Visit 2. Participants will participate in the same type of task inside the MRI scanner, while the study staff measures reaction time and psychophysiological responding and brain activation. Participants will view the same images he or she did previously, and may experience the same aversive stimulus as during Visit 2. Participants will again be asked to rate how much they expect to experience the aversive stimulus after each image and will also be asked to report their level of anxiety on a scale from 0 to 100.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Able to give informed consent
* Physically and neurologically healthy [confirmed by a comprehensive medical history]
* Age between 21-45 years old
* Right-handed

Inclusion Criteria for Participants with PTSD:

* Current PTSD diagnosis [related to civilian trauma]

Inclusion Criteria for Trauma-Exposed Participants without PTSD:

* Experience with a civilian trauma without a PTSD diagnosis
* Free of a lifetime Axis I or Axis II diagnosis

Inclusion Criteria for Non-Trauma-Exposed Healthy Participants:

* Free of a lifetime Axis I or Axis II diagnosis

Exclusion Criteria for All Participants:

* Clinically significant medical or neurological condition
* Less than a high school education
* Lack of fluency in English
* Night shift work
* Currently pregnant; planning pregnancy; or lactating
* Unwilling/unable to sign informed consent document
* Inability to tolerate small, enclosed spaces without anxiety (e.g. claustrophobia)
* Left-handed
* Presence of ferrous-containing metals within the body (e.g., aneurysm clips, shrapnel/retained particles)
* Under 21 or over 45 years of age
* Anticipation of a required drug test in the 4 weeks following study participation
* Positive urine drug screen and/or alcohol breathalyzer
* Current or past allergic or adverse reaction or known sensitivity to cannabinoid-like substances [dronabinol/marijuana/cannabis/thc, cannabinoid oil, sesame oil, gelatin, glycerin, and titanium dioxide]
* Participation in an experiment involving white noise bursts or shocks in the last 6 months

Exclusion Criteria for Participants with PTSD:

* Primary comorbid anxiety disorder (defined by which disorder was the more debilitating and clinically salient)
* Life history of bipolar disorder, schizophrenia, or presence of an organic mental syndrome, mental retardation, or pervasive developmental disorder
* Current or in the past 6 months alcohol/drug abuse of dependence
* Current or in the past 6 months major depressive disorder
* Current suicidal ideation
* Diagnosis of an Axis II personality disorder
* Concomitant treatments with psychotropic/psychoactive medication [including beta-adrenergic blockers, selective serotonin reuptake inhibitor (SSRI), benzodiazepines, tricyclic or monoamine oxidase inhibitor (MAOI) antidepressants, lithium, antiepileptic/anticonvulsants, neuroleptics/antipsychotics, etc.) or in the past two weeks [8 weeks for fluoxetine and 4 weeks for MAOIs) before screening (Visit 1)
* currently receiving exposure-based therapy for PTSD

Exclusion Criteria for Trauma-Exposed Participants without PTSD and Non-Trauma Exposed Healthy Participants:

* Current or past Axis I psychiatric disorder [including alcohol/substance abuse of dependence disorder]

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine A. Rabinak, PhD, Principal Investigator — Wayne State University
Locations (1):
- Eugene Applebaum College of Pharmacy and Health Sciences, Detroit, Michigan, United States

REFERENCES:
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873

RESULTS

PARTICIPANT FLOW:
Groups:
- PTSD-dronabinol: Trauma exposed individuals with PTSD that received a one-time oral dose of dronabinol (7.5mg)
- PTSD-placebo: Trauma exposed individuals with PTSD that received a one-time oral dose of placebo
- TEC-dronabinol: Trauma exposed individuals without PTSD that received a one-time oral dose of dronabinol (7.5mg)
- TEC-placebo: Trauma exposed individuals without PTSD that received a one-time oral dose of placebo
- HC-dronabinol: Non-trauma exposed individuals that received a one-time oral dose of dronabinol (7.5mg)
- HC-placebo: Non-trauma exposed individuals that received a one-time oral dose of placebo
Period: Overall Study
Arm/Group | PTSD-dronabinol | PTSD-placebo | TEC-dronabinol | TEC-placebo | HC-dronabinol | HC-placebo
Started | 13 | 10 | 18 | 17 | 14 | 14
Completed | 12 | 10 | 15 | 15 | 14 | 12
Not Completed | 1 | 0 | 3 | 2 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PTSD-dronabinol: Trauma-exposed individuals with PTSD that received a one-time oral dose of dronabinol (7.5mg)
- PTSD-placebo: Trauma-exposed individuals with PTSD that received a one-time oral dose of placebo
- TEC-dronabinol: Trauma-exposed individuals without PTSD that received a one-time oral dose of dronabinol (7.5mg)
- TEC-placebo: Trauma-exposed individuals without PTSD that received a one-time oral dose of placebo
- HC-dronabinol: Non-trauma-exposed individuals that received a one-time oral dose of dronabinol (7.5mg)
- HC-placebo: Non-trauma-exposed individuals that received a one-time oral dose of placebo
- Total: Total of all reporting groups
Arm/Group | PTSD-dronabinol | PTSD-placebo | TEC-dronabinol | TEC-placebo | HC-dronabinol | HC-placebo | Total
Number analyzed (Participants) | 13 | 10 | 18 | 17 | 14 | 14 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 18 | 17 | 14 | 14 | 86
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.69 (4.91) | 23.40 (2.91) | 28.94 (7.50) | 26.59 (6.83) | 24.29 (2.46) | 25.79 (4.77) | 26.07 (5.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 6 | 11 | 6 | 3 | 43
  Male | 2 | 4 | 12 | 6 | 8 | 11 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 1 | 1 | 0 | 2 | 7
  Not Hispanic or Latino | 10 | 10 | 17 | 16 | 14 | 12 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 1 | 3 | 5 | 6 | 4 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 6 | 4 | 0 | 3 | 18
  White | 8 | 6 | 8 | 6 | 8 | 7 | 43
  More than one race | 1 | 1 | 0 | 1 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 18 | 17 | 14 | 14 | 86

OUTCOME MEASURES:

1. Primary Outcome: Brain Measures
Description: Mean functional magnetic resonance imaging (fMRI) BOLD activation extracted from each region of interests [amygdala; ventromedial prefrontal cortex; hippocampus] for each stimulus type (CS+E, CS+U, CS-). The units of BOLD values are expressed as arbitrary units.
Time Frame: Brain measures are collected on Visit 3, 14 days from baseline (Visit 1) and Visit 4, 15 days from baseline (Visit 1), for approximately 1.5 hours each day
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | PTSD-dronabinol | PTSD-placebo | TEC-dronabinol | TEC-placebo | HC-dronabinol | HC-placebo
Number analyzed (Participants) | 12 | 10 | 15 | 15 | 14 | 12
arbitrary units
  Extinction Learning CS+E Amygdala- Visit 3 | -0.08 (0.23) | 0.27 (0.27) | 0.02 (0.21) | 0.03 (0.27) | -0.05 (0.28) | -0.09 (0.30)
  Extinction Learning CS+E Hippocampus- Visit 3 | -0.06 (0.12) | -0.03 (0.13) | -0.07 (0.09) | -0.06 (0.15) | -0.05 (0.08) | -0.14 (0.23)
  Extinction Learning CS+E vmPFC- Visit 3 | -0.11 (0.15) | -0.22 (0.19) | -0.12 (0.21) | -0.14 (0.19) | -0.18 (0.16) | -0.21 (0.18)
  Extinction Learning CS- Amygdala- Visit 3 | -0.01 (0.34) | 0.19 (0.22) | 0.07 (0.23) | 0.04 (0.22) | 0.02 (0.28) | -0.07 (0.31)
  Extinction Learning CS- Hippocampus- Visit 3 | -0.04 (0.19) | -0.05 (0.11) | -0.04 (0.16) | -0.01 (0.12) | -0.07 (0.16) | -0.14 (0.20)
  Extinction Learning CS- vmPFC- Visit 3 | -0.10 (0.16) | -0.23 (0.13) | -0.16 (0.19) | -0.10 (0.13) | -0.17 (0.23) | -0.17 (0.21)
  Recall CS+E Amygdala- Visit 4 | 0.20 (0.24) | 0.10 (0.33) | 0.11 (0.19) | 0.03 (0.32) | 0.01 (0.12) | -0.01 (0.33)
  Recall CS+E Hippocampus-Visit 4 | 0.05 (0.12) | -0.02 (0.15) | 0.04 (0.13) | 0.01 (0.18) | 0.0 (0.17) | 0.0 (0.26)
  Recall CS+E vmPFC-Visit 4 | -0.19 (0.26) | -0.06 (0.12) | -0.08 (0.14) | -0.14 (0.26) | -0.11 (0.22) | -0.19 (0.28)
  Recall CS- Amygdala-Visit 4 | 0.14 (0.36) | 0.18 (0.41) | 0.01 (0.20) | -0.02 (0.20) | 0.16 (0.15) | 0.20 (0.31)
  Recall CS- Hippocampus-Visit 4 | 0.02 (0.20) | 0.0 (0.23) | -0.04 (0.07) | -0.02 (0.12) | 0.04 (0.14) | 0.09 (0.19)
  Recall CS- vmPFC-Visit 4 | -0.15 (0.19) | -0.05 (0.16) | -0.20 (0.21) | -0.16 (0.19) | -0.12 (0.18) | -0.10 (0.19)
  Recall CS+U Amygdala-Visit 4 | 0.12 (0.23) | 0.14 (0.20) | 0.14 (0.24) | -0.06 (0.24) | 0.09 (0.19) | 0.06 (0.21)
  Recall CS+U Hippocampus-Visit 4 | -0.04 (0.11) | -0.05 (0.15) | -0.02 (0.11) | -0.05 (0.10) | 0 (0.19) | 0 (0.15)
  Recall CS+U vmPFC-Visit 4 | -0.18 (0.25) | -0.08 (0.21) | -0.24 (0.23) | -0.20 (0.17) | -0.14 (0.21) | -0.16 (0.28)
  Renewal CS+E Amygdala-Visit 4 | 0.16 (0.21) | 0.19 (0.43) | 0.13 (0.23) | 0.06 (0.24) | 0.10 (0.17) | 0.07 (0.32)
  Renewal CS+E Hippocampus- Visit 4 | 0.11 (0.08) | 0.06 (0.25) | 0.04 (0.07) | 0.04 (0.13) | 0.03 (0.18) | 0.04 (0.15)
  Renewal CS+E vmPFC- Visit 4 | 0.0 (0.20) | -0.09 (0.22) | -0.14 (0.18) | -0.12 (0.29) | -0.08 (0.2) | -0.08 (0.19)
  Renewal CS- Amygdala- Visit 4 | 0.04 (0.15) | 0.25 (0.36) | -0.10 (0.21) | -0.02 (0.37) | 0.04 (0.18) | 0.19 (0.31)
  Renewal CS- Hippocampus-Visit 4 | 0.02 (0.12) | 0.06 (0.19) | -0.03 (0.08) | 0.01 (0.22) | 0.06 (0.08) | 0.05 (0.16)
  Renewal CS- vmPFC-Visit 4 | -0.10 (0.26) | -0.05 (0.20) | -0.14 (0.22) | -0.15 (0.20) | -0.10 (0.20) | -0.12 (0.25)
  Renewal CS+U Amygdala-Visit 4 | 0.05 (0.18) | 0.22 (0.31) | 0.09 (0.22) | 0.09 (0.31) | 0.03 (0.32) | -0.04 (0.30)
  Renewal CS+U Hippocampus-Visit 4 | 0.01 (0.13) | 0.06 (0.16) | 0.09 (0.11) | 0.06 (0.11) | -0.01 (0.16) | -0.05 (0.21)
  Renewal CS+U vmPFC-Visit 4 | -0.20 (0.22) | -0.07 (0.20) | -0.04 (0.19) | -0.12 (0.19) | -0.15 (0.17) | -0.18 (0.20)
Statistical Analysis 1: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Extinction Learning CS+E Amygdala- Visit 3' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p > 0.05, ANOVA — RM-ANOVA. Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 2: Comparison: PTSD-placebo vs TEC-placebo vs HC-placebo; This analysis corresponds to the row 'Extinction Learning CS+E Hippocampus- Visit 3' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p = 0.041, ANOVA — Repeated-measures ANOVA (SPM12, ROI small-volume corrected). Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 3: Comparison: PTSD-dronabinol vs TEC-dronabinol; This analysis corresponds to the row 'Extinction Learning CS+E vmPFC- Visit 3' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p = 0.040, ANOVA — Repeated-measures ANOVA (SPM12, ROI small-volume corrected). Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 4: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Extinction Learning CS- Amygdala- Visit 3' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p > 0.05, ANOVA — RM-ANOVA. Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 5: Comparison: PTSD-placebo vs TEC-placebo vs HC-placebo; This analysis corresponds to the row 'Extinction Learning CS- Hippocampus- Visit 3' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p = 0.041, ANOVA — Repeated-measures ANOVA (SPM12, ROI small-volume corrected). Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 6: Comparison: PTSD-dronabinol vs TEC-dronabinol; This analysis corresponds to the row 'Extinction Learning CS- vmPFC- Visit 3' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p = 0.040, ANOVA — Repeated-measures ANOVA (SPM12, ROI small-volume corrected). Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus time factors
Statistical Analysis 7: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Recall CS+E Amygdala- Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p > 0.05, ANOVA — RM-ANOVA. Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 8: Comparison: PTSD-dronabinol vs TEC-dronabinol vs HC-dronabinol; This analysis corresponds to the row 'Recall CS+E Hippocampus-Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p = 0.027, ANOVA — Repeated-measures ANOVA (SPM12, ROI small-volume corrected). Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 9: Comparison: PTSD-placebo vs TEC-placebo vs HC-placebo; This analysis corresponds to the row 'Recall CS+E vmPFC-Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p = 0.019, ANOVA — Repeated-measures ANOVA (SPM12, ROI small-volume corrected). Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 10: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Recall CS- Amygdala-Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p > 0.05, ANOVA — RM-ANOVA. Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 11: Comparison: PTSD-dronabinol vs TEC-dronabinol vs HC-dronabinol; This analysis corresponds to the row 'Recall CS- Hippocampus-Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p = 0.027, ANOVA — Repeated-measures ANOVA (SPM12, ROI small-volume corrected). Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 12: Comparison: PTSD-placebo vs TEC-placebo vs HC-placebo; This analysis corresponds to the row 'Recall CS- vmPFC-Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p = 0.019, ANOVA — Repeated-measures ANOVA (SPM12, ROI small-volume corrected). Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 13: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Recall CS+U Amygdala-Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p > 0.05, ANOVA — RM-ANOVA. Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 14: Comparison: PTSD-dronabinol vs TEC-dronabinol vs HC-dronabinol; This analysis corresponds to the row 'Recall CS+U Hippocampus-Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p = 0.027, ANOVA — Repeated-measures ANOVA (SPM12, ROI small-volume corrected). Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 15: Comparison: PTSD-placebo vs TEC-placebo vs HC-placebo; This analysis corresponds to the row 'Recall CS+U vmPFC-Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p = 0.019, ANOVA — Repeated-measures ANOVA (SPM12, ROI small-volume corrected). Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 16: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal CS+E Amygdala-Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p > 0.05, ANOVA — RM-ANOVA. Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 17: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal CS+E Hippocampus- Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p > 0.05, ANOVA — RM-ANOVA. Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 18: Comparison: PTSD-dronabinol vs TEC-dronabinol vs HC-dronabinol; This analysis corresponds to the row 'Renewal CS+E vmPFC- Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p = 0.025, ANOVA — Repeated-measures ANOVA (SPM12, ROI small-volume corrected). Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 19: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal CS- Amygdala- Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p > 0.05, ANOVA — RM-ANOVA. Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 20: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal CS- Hippocampus-Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p > 0.05, ANOVA — RM-ANOVA. Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 21: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal CS- vmPFC-Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p > 0.05, ANOVA — RM-ANOVA. Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 22: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal CS+U Amygdala-Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p > 0.05, ANOVA — RM-ANOVA. Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 23: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal CS+U Hippocampus-Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p > 0.05, ANOVA — RM-ANOVA. Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors
Statistical Analysis 24: Comparison: PTSD-dronabinol vs TEC-dronabinol vs HC-dronabinol; This analysis corresponds to the row 'Renewal CS+U vmPFC-Visit 4' in the Brain Measures outcome table. RM-ANOVA including stimulus (CS+E, CS-, CS+U); Test type: Superiority; p = 0.025, ANOVA — Repeated-measures ANOVA (SPM12, ROI small-volume corrected). Significance threshold p<0.05, FWE-corrected; RM-ANOVA with group and stimulus factors

2. Primary Outcome: Expectancy Ratings
Description: To assess the expected likelihood that an aversive cue (e.g. noise burst) will occur or not based on the CS shown on the screen. Participants rate their expectancy of the aversive cue using a button box on a scale from 1 to 3 [1 = certain that the aversive cue will be presented (Yes); 2 = certain that the aversive cue will not be presented (No); 3 = uncertain whether the aversive cue will be presented (I don't know)]. Counts of "yes", "no", and "I don't know" are collected on the first (early) trial of the CS and the last (late) trial of the CS.
Time Frame: Collected on Visit 2, 13 days from baseline (Visit 1), Visit 3, 14 days from baseline (Visit 1), and Visit 4, 15 days from baseline, during the task. Each day the task lasted approximately 20 minutes.
Population: The number analyzed in each row may differ from the overall number analyzed due to missing data.
Measure: Count of Participants; unit: Participants
Groups:
- HC-placebo: Non-trauma-exposed individuals with PTSD that received a one-time oral dose of placebo
Arm/Group | PTSD-dronabinol | PTSD-placebo | TEC-dronabinol | TEC-placebo | HC-dronabinol | HC-placebo
Number analyzed (Participants) | 12 | 10 | 15 | 15 | 14 | 12
Participants
  Acquisition CS+E Early- Visit 2: number analyzed (Participants) | 7 | 10 | 12 | 14 | 12 | 12
  Acquisition CS+E Early- Visit 2: No | 1 | 3 | 4 | 2 | 3 | 4
  Acquisition CS+E Early- Visit 2: I don't know | 0 | 0 | 1 | 0 | 0 | 0
  Acquisition CS+E Early- Visit 2: Yes | 6 | 7 | 7 | 12 | 9 | 8
  Acquisition CS+U Early- Visit 2: number analyzed (Participants) | 7 | 10 | 12 | 14 | 12 | 12
  Acquisition CS+U Early- Visit 2: No | 2 | 3 | 3 | 5 | 2 | 5
  Acquisition CS+U Early- Visit 2: I don't know | 0 | 1 | 1 | 0 | 0 | 2
  Acquisition CS+U Early- Visit 2: Yes | 5 | 6 | 8 | 9 | 10 | 5
  Acquisition CS-Early- Visit 2: number analyzed (Participants) | 7 | 10 | 12 | 14 | 12 | 12
  Acquisition CS-Early- Visit 2: No | 5 | 6 | 6 | 6 | 11 | 8
  Acquisition CS-Early- Visit 2: I don't know | 0 | 0 | 3 | 4 | 0 | 0
  Acquisition CS-Early- Visit 2: Yes | 2 | 4 | 3 | 4 | 1 | 4
  Acquisition CS+E Late- Visit 2: number analyzed (Participants) | 7 | 10 | 12 | 14 | 12 | 12
  Acquisition CS+E Late- Visit 2: No | 1 | 4 | 5 | 1 | 3 | 2
  Acquisition CS+E Late- Visit 2: I don't know | 0 | 0 | 0 | 2 | 1 | 1
  Acquisition CS+E Late- Visit 2: Yes | 6 | 6 | 7 | 11 | 8 | 9
  Acquisition CS+U Late- Visit 2: number analyzed (Participants) | 7 | 10 | 12 | 13 | 12 | 12
  Acquisition CS+U Late- Visit 2: No | 3 | 3 | 3 | 1 | 3 | 1
  Acquisition CS+U Late- Visit 2: I don't know | 0 | 1 | 2 | 1 | 4 | 1
  Acquisition CS+U Late- Visit 2: Yes | 4 | 6 | 7 | 11 | 5 | 10
  Acquisition CS- Late- Visit 2: number analyzed (Participants) | 7 | 10 | 12 | 14 | 12 | 12
  Acquisition CS- Late- Visit 2: No | 7 | 8 | 8 | 13 | 11 | 10
  Acquisition CS- Late- Visit 2: I don't know | 0 | 1 | 1 | 0 | 0 | 1
  Acquisition CS- Late- Visit 2: Yes | 0 | 1 | 3 | 1 | 1 | 1
  Extinction CS+E Early- Visit 3: number analyzed (Participants) | 9 | 10 | 11 | 14 | 12 | 12
  Extinction CS+E Early- Visit 3: No | 0 | 1 | 3 | 3 | 2 | 4
  Extinction CS+E Early- Visit 3: I don't know | 2 | 4 | 1 | 2 | 2 | 0
  Extinction CS+E Early- Visit 3: Yes | 7 | 5 | 7 | 9 | 8 | 8
  Extinction CS- Early- Visit 3: number analyzed (Participants) | 9 | 10 | 11 | 14 | 12 | 12
  Extinction CS- Early- Visit 3: No | 5 | 3 | 3 | 6 | 4 | 6
  Extinction CS- Early- Visit 3: I don't know | 1 | 6 | 5 | 4 | 5 | 0
  Extinction CS- Early- Visit 3: Yes | 3 | 1 | 3 | 4 | 3 | 6
  Extinction CS+E Late-Visit 3: number analyzed (Participants) | 9 | 10 | 11 | 14 | 13 | 12
  Extinction CS+E Late-Visit 3: No | 6 | 7 | 7 | 6 | 10 | 5
  Extinction CS+E Late-Visit 3: I don't know | 0 | 0 | 1 | 2 | 1 | 0
  Extinction CS+E Late-Visit 3: Yes | 3 | 3 | 3 | 6 | 2 | 7
  Extinction CS- Late- Visit 3: number analyzed (Participants) | 8 | 10 | 11 | 14 | 13 | 12
  Extinction CS- Late- Visit 3: No | 5 | 9 | 9 | 13 | 9 | 6
  Extinction CS- Late- Visit 3: I don't know | 2 | 0 | 0 | 1 | 1 | 0
  Extinction CS- Late- Visit 3: Yes | 1 | 1 | 2 | 0 | 3 | 6
  Recall CS+E Early-Visit 4: number analyzed (Participants) | 9 | 10 | 12 | 14 | 13 | 12
  Recall CS+E Early-Visit 4: No | 3 | 4 | 5 | 5 | 3 | 5
  Recall CS+E Early-Visit 4: I don't know | 3 | 3 | 2 | 2 | 4 | 1
  Recall CS+E Early-Visit 4: Yes | 3 | 3 | 5 | 7 | 6 | 6
  Recall CS+U Early-Visit 4: number analyzed (Participants) | 9 | 10 | 12 | 14 | 13 | 12
  Recall CS+U Early-Visit 4: No | 4 | 1 | 5 | 4 | 4 | 5
  Recall CS+U Early-Visit 4: I don't know | 4 | 3 | 2 | 5 | 5 | 1
  Recall CS+U Early-Visit 4: Yes | 1 | 6 | 5 | 5 | 4 | 6
  Recall CS- Early-Visit 4: number analyzed (Participants) | 9 | 10 | 11 | 14 | 13 | 12
  Recall CS- Early-Visit 4: No | 3 | 6 | 7 | 7 | 8 | 7
  Recall CS- Early-Visit 4: I don't know | 4 | 3 | 4 | 2 | 1 | 0
  Recall CS- Early-Visit 4: Yes | 2 | 1 | 0 | 5 | 4 | 5
  Recall CS+E Late-Visit 4: number analyzed (Participants) | 9 | 10 | 11 | 14 | 12 | 12
  Recall CS+E Late-Visit 4: No | 7 | 8 | 9 | 7 | 7 | 7
  Recall CS+E Late-Visit 4: I don't know | 1 | 0 | 0 | 3 | 0 | 0
  Recall CS+E Late-Visit 4: Yes | 1 | 2 | 2 | 4 | 5 | 5
  Recall CS+U Late-Visit 4: number analyzed (Participants) | 9 | 10 | 12 | 13 | 12 | 10
  Recall CS+U Late-Visit 4: No | 4 | 5 | 11 | 8 | 8 | 4
  Recall CS+U Late-Visit 4: I don't know | 2 | 0 | 0 | 1 | 1 | 0
  Recall CS+U Late-Visit 4: Yes | 3 | 5 | 1 | 4 | 3 | 6
  Recall CS- Late-Visit 4: number analyzed (Participants) | 9 | 9 | 11 | 13 | 13 | 12
  Recall CS- Late-Visit 4: No | 6 | 8 | 9 | 8 | 9 | 6
  Recall CS- Late-Visit 4: I don't know | 2 | 0 | 1 | 4 | 0 | 0
  Recall CS- Late-Visit 4: Yes | 1 | 1 | 1 | 1 | 4 | 6
  Renewal CS+E Early-Visit 4: number analyzed (Participants) | 9 | 10 | 12 | 14 | 13 | 12
  Renewal CS+E Early-Visit 4: No | 4 | 2 | 3 | 3 | 3 | 6
  Renewal CS+E Early-Visit 4: I don't know | 2 | 2 | 2 | 5 | 4 | 1
  Renewal CS+E Early-Visit 4: Yes | 3 | 6 | 7 | 6 | 6 | 5
  Renewal CS+U Early-Visit 4: number analyzed (Participants) | 9 | 10 | 12 | 14 | 12 | 12
  Renewal CS+U Early-Visit 4: No | 4 | 2 | 8 | 3 | 4 | 5
  Renewal CS+U Early-Visit 4: I don't know | 1 | 2 | 3 | 6 | 5 | 2
  Renewal CS+U Early-Visit 4: Yes | 4 | 6 | 1 | 5 | 3 | 5
  Renewal CS- Early-Visit 4: number analyzed (Participants) | 9 | 9 | 12 | 14 | 13 | 12
  Renewal CS- Early-Visit 4: No | 8 | 7 | 7 | 8 | 11 | 7
  Renewal CS- Early-Visit 4: I don't know | 1 | 2 | 3 | 2 | 0 | 0
  Renewal CS- Early-Visit 4: Yes | 0 | 0 | 2 | 4 | 2 | 5
  Renewal CS+E Late-Visit 4: number analyzed (Participants) | 9 | 10 | 12 | 13 | 13 | 11
  Renewal CS+E Late-Visit 4: No | 7 | 8 | 10 | 5 | 8 | 6
  Renewal CS+E Late-Visit 4: I don't know | 1 | 0 | 0 | 2 | 1 | 0
  Renewal CS+E Late-Visit 4: Yes | 1 | 2 | 2 | 6 | 4 | 5
  Renewal CS+U Late-Visit 4: number analyzed (Participants) | 9 | 10 | 11 | 13 | 12 | 12
  Renewal CS+U Late-Visit 4: No | 5 | 5 | 10 | 6 | 6 | 6
  Renewal CS+U Late-Visit 4: I don't know | 2 | 0 | 0 | 3 | 2 | 0
  Renewal CS+U Late-Visit 4: Yes | 2 | 5 | 1 | 4 | 4 | 6
  Renewal CS- Late-Visit 4: number analyzed (Participants) | 8 | 10 | 11 | 13 | 13 | 12
  Renewal CS- Late-Visit 4: No | 6 | 9 | 10 | 9 | 11 | 8
  Renewal CS- Late-Visit 4: I don't know | 1 | 1 | 1 | 2 | 1 | 0
  Renewal CS- Late-Visit 4: Yes | 1 | 0 | 0 | 2 | 1 | 4
Statistical Analysis 1: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Acquisition CS+E Early- Visit 2' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 2: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Acquisition CS+U Early- Visit 2' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 3: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Acquisition CS-Early- Visit 2' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 4: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Acquisition CS+E Late- Visit 2' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 5: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Acquisition CS+U Late- Visit 2' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 6: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Acquisition CS- Late- Visit 2' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 7: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Extinction CS+E Early- Visit 3' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 8: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Extinction CS- Early- Visit 3' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 9: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Extinction CS+E Late-Visit 3' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 10: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Extinction CS- Late- Visit 3' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p = 0.04, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 11: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Recall CS+E Early-Visit 4' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 12: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Recall CS+U Early-Visit 4' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 13: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Recall CS- Early-Visit 4' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 14: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Recall CS+E Late-Visit 4' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 15: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Recall CS+U Late-Visit 4' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 16: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Recall CS- Late-Visit 4' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p = 0.033, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 17: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal CS+E Early-Visit 4' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 18: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal CS+U Early-Visit 4' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 19: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal CS- Early-Visit 4' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 20: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal CS+E Late-Visit 4' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 21: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal CS+U Late-Visit 4' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10
Statistical Analysis 22: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal CS- Late-Visit 4' in the Expectancy Ratings outcome table. Chi-square test comparing distribution of Yes/No/I don't know responses across 6 groups; Test type: Superiority; p > 0.05, Chi-squared — Chi-square test of independence; significance threshold p<0.05; 3 (response categories) × 6 (groups) contingency table; df=10

3. Secondary Outcome: Subjective Units of Distress (SUDS)
Description: Subjective Units of Distress (SUDS): used to measure fear ratings/"subjective" anxiety on a scale from 0-10; taken at three time points throughout the tasks: before the task begins, in the middle of the task, and at the end of the task. A rating of "0" means no anxiety and a ratings of "10" means worst anxiety ever experienced.
Time Frame: SUDS ratings are collected at Visit 3 (Day 14 from baseline) and Visit 4 (Day 15 from baseline), at three timepoints per visit: before the task (Pre), midpoint (Mid), and after the task (Post), each averaged over ~1 minute.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PTSD-dronabinol | PTSD-placebo | TEC-dronabinol | TEC-placebo | HC-dronabinol | HC-placebo
Number analyzed (Participants) | 12 | 10 | 15 | 15 | 14 | 12
score on a scale
  Extinction Learning Pre- Visit 3 | 3.44 (2.7) | 2.5 (1.58) | 2.83 (1.95) | 1.79 (2.29) | 3.15 (2.03) | 1.92 (1.32)
  Extinction Learning Mid-Visit 3 | 4.22 (2.82) | 2.90 (2.38) | 3.50 (2.54) | 1.50 (1.56) | 3.00 (2.58) | 2.23 (2.20)
  Extinction Learning Post-Visit 3 | 3.56 (2.55) | 2.20 (1.87) | 2.75 (2.42) | 1.64 (2.06) | 3.23 (2.52) | 2.31 (2.39)
  Recall Pre-Visit 4 | 1.22 (0.97) | 2.00 (2.26) | 0.92 (1.44) | 0.50 (1.40) | 1.46 (1.94) | 1.00 (1.47)
  Recall Mid-Visit 4 | 2.00 (1.87) | 2.20 (1.99) | 1.42 (2.31) | 0.64 (1.39) | 1.46 (1.76) | 1.08 (1.75)
  Recall Post-Visit 4 | 1.56 (1.81) | 1.70 (2.21) | 1.25 (2.26) | 1.21 (1.53) | 1.38 (1.76) | 1.77 (1.76)
  Renewal Pre-Visit 4 | 1.56 (1.13) | 2.10 (2.23) | 1.25 (2.01) | 0.93 (1.00) | 1.46 (1.56) | 1.54 (2.18)
  Renewal Mid-Visit 4 | 1.67 (1.12) | 1.80 (2.30) | 1.25 (1.76) | 1.29 (1.68) | 1.54 (1.51) | 1.46 (2.03)
  Renewal Post-Visit 4 | 1.89 (1.54) | 2.00 (3.02) | 1.17 (1.70) | 1.50 (2.14) | 1.38 (1.33) | 1.62 (2.02)
Statistical Analysis 1: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Extinction Learning Pre- Visit 3' in the SUDS outcome table. ANOVA comparing mean SUDS ratings across 6 groups at the specified phase/timepoint; Test type: Superiority; p > 0.05, ANOVA — Significance threshold p<0.05; Group factor at specified phase/timepoint
Statistical Analysis 2: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Extinction Learning Mid-Visit 3' in the SUDS outcome table. ANOVA comparing mean SUDS ratings across 6 groups at the specified phase/timepoint; Test type: Superiority; p > 0.05, ANOVA — Significance threshold p<0.05; Group factor at specified phase/timepoint
Statistical Analysis 3: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Extinction Learning Post-Visit 3' in the SUDS outcome table. ANOVA comparing mean SUDS ratings across 6 groups at the specified phase/timepoint; Test type: Superiority; p > 0.05, ANOVA — Significance threshold p<0.05; Group factor at specified phase/timepoint
Statistical Analysis 4: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Recall Pre-Visit 4' in the SUDS outcome table. ANOVA comparing mean SUDS ratings across 6 groups at the specified phase/timepoint; Test type: Superiority; p > 0.05, ANOVA — Significance threshold p<0.05; Group factor at specified phase/timepoint
Statistical Analysis 5: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Recall Mid-Visit 4' in the SUDS outcome table. ANOVA comparing mean SUDS ratings across 6 groups at the specified phase/timepoint; Test type: Superiority; p > 0.05, ANOVA — Significance threshold p<0.05; Group factor at specified phase/timepoint
Statistical Analysis 6: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Recall Post-Visit 4' in the SUDS outcome table. ANOVA comparing mean SUDS ratings across 6 groups at the specified phase/timepoint; Test type: Superiority; p > 0.05, ANOVA — Significance threshold p<0.05; Group factor at specified phase/timepoint
Statistical Analysis 7: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal Pre-Visit 4' in the SUDS outcome table. ANOVA comparing mean SUDS ratings across 6 groups at the specified phase/timepoint; Test type: Superiority; p > 0.05, ANOVA — Significance threshold p<0.05; Group factor at specified phase/timepoint
Statistical Analysis 8: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal Mid-Visit 4' in the SUDS outcome table. ANOVA comparing mean SUDS ratings across 6 groups at the specified phase/timepoint; Test type: Superiority; p > 0.05, ANOVA — Significance threshold p<0.05; Group factor at specified phase/timepoint
Statistical Analysis 9: Comparison: PTSD-dronabinol vs PTSD-placebo vs TEC-dronabinol vs TEC-placebo vs HC-dronabinol vs HC-placebo; This analysis corresponds to the row 'Renewal Post-Visit 4' in the SUDS outcome table. ANOVA comparing mean SUDS ratings across 6 groups at the specified phase/timepoint; Test type: Superiority; p > 0.05, ANOVA — Significance threshold p<0.05; Group factor at specified phase/timepoint

ADVERSE EVENTS:
Time Frame: Adverse event data was collected starting when a participant was classified as enrolled in the study and continued until they completed all study visits, which was no more than 3 weeks.
Arm/Group | PTSD-dronabinol | PTSD-placebo | TEC-dronabinol | TEC-placebo | HC-dronabinol | HC-placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10 | 0/18 | 0/17 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10 | 0/18 | 0/17 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/10 | 0/18 | 0/17 | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT02069366/Prot_SAP_000.pdf